CLINICAL TRIAL: NCT03985605
Title: Therapeutic Drug Monitoring of Antiinfectives for Patients With Severe Illness
Brief Title: Therapeutic Drug Monitoring of Antiinfectives for Patients With Severe Illness = TAPSI
Acronym: TAPSI
Status: Completed | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Michael Zoller MD, Principal Investigator, Ludwig-Maximilians - University of Munich
Other Study IDs: LMU 18-578
Record Dates: First submitted 2019-05-27; First posted 2019-06-14 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Infection, Bacterial
Keywords: TDM; Routine; intensive care patients
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Therapeutic drug monitoring of antiinfectives in intensive care patients is an usual research topic of the last years. Based on research result, which have shown subtherapeutic plasma concentrations of antibiotics, a routines therapeutic drug monitoring for β-lactam-antibiotics was implemented in January 2018 at Clinic for Anesthesiology at University Hospital, LMU Munich, Germany. This study is an prospective evaluation of these TDM-program.

DETAILED DESCRIPTION:
Bacterial infections are associated with high mortality in intensive care patients. Antibiotic therapy is the only causal opportunity to treat those infections. Pharmacokinetic and -dynamic changes in critically ill patients lead to unpredictable plasma concentrations of the applied drugs. Research results of the last years with many quantified plasma concentrations in subtherapeutic levels yield to the recommendation of the Paul-Ehrlich-Society for an routines therapeutic drug monitoring of antibiotics in intensive care patients. These was implemented in January 2018 at Clinic for Anesthesiology at University Hospital, LMU Munich, Germany for all intensive care patients as a routines procedure. The introduced study is a prospective evaluation of the TDM-program with regard to improvement opportunity, influencing factors and parallels to other studies.

ELIGIBILITY:
Inclusion Criteria:

* routines TDM of antiinfectives

Exclusion Criteria:

* TDM is not available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill intensive care patients who were included in the routines TDM-program since January 2018.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Incidence of subtherapeutic antiinfective concentrations | four years
  Number of subtherapeutic concentrations from different antiinfectives in critically ill patients
Correlation of meropenem concentration in serum to the concentration in brain fluid | during the treatment with an external ventricular drainage
  The concentration of meropenem in the brain fluid of 30 patients with an external ventricular drainage will be correlated to their serum concentration
Subtherapeutic antiinfective concentrations during hemoadsorption | during hemoadsorption treatment
  Subtherapeutic concentrations of antiinfectives in serum during hemoadsorption treatment

SECONDARY OUTCOMES:
28-day mortality of patients with therapeutic drug monitoring of antiinfectives | during intensive care treatment
  Correlation of antiinfective concentrations in serum to 28-day mortality
ICU-free days of patients with therapeutic drug monitoring of antiinfectives | during intensive care treatment
  Correlation of antiinfective concentrations in serum to ICU-free days to day 28
Sofa-score course of patients with therapeutic drug monitoring of antiinfectives | during the treatment with the antiinfectives
  Correlation of antiinfective concentrations in serum to sofa-score
Time course of Interleukin-6 in patients with therapeutic drug monitoring of antiinfectives | during the treatment with the antiinfectives
  Correlation of antiinfective concentrations to Interleukin-6 in critically ill patients
Time course of CRP in patients with therapeutic drug monitoring of antiinfectives | during the treatment with the antiinfectives
  Correlation of antiinfective concentrations to CRP in critically ill patients

CONTACTS AND LOCATIONS:
Overall Officials: Bruegel Mathias, Dr. med., Principal Investigator — Institute of Laboratory Medicine of the University Hospital of Munich; Liebchen Uwe, Dr.med., Study Chair — Department of Anaesthesiology of the University Hospital of Munich; Ines Schroeder, Dr.med., Study Chair — Department of Anaesthesiology of the University Hospital of Munich; Paal Michael, Dr.rer.nat., Study Chair — Institute of Laboratory Medicine of the University Hospital of Munich; Bernhard Zwissler, Prof.Dr.med., Study Director — Department of Anaesthesiology of the University Hospital of Munich; Daniel Teupser, Prof.Dr.med., Study Director — Institute of Laboratory Medicine of the University Hospital of Munich; Lesca Holdt, Prof.Dr.med., Study Chair — Institute of Laboratory Medicine of the University Hospital of Munich; Michael Vogeser, Prof.Dr.med., Study Chair — Institute of Laboratory Medicine of the University Hospital of Munich; Eike Speck, Study Chair — Department of Anaesthesiology of the University Hospital of Munich; Michael Irlbeck, PD.Dr.med., Study Chair — Department of Anaesthesiology of the University Hospital of Munich; Thomas Weig, PD.Dr.med., Study Chair — Department of Anaesthesiology of the University Hospital of Munich
Locations (1):
- Department of Anaesthesiology of the University Hospital of Munich, Munich, Germany

IPD SHARING:
Plan to Share IPD: No
sharing individual participant data is restricted by EU General Data Protection Regulation (GDPR)

REFERENCES:
- [Derived] Weber F, Scharf C, Aulin LBS, Weinelt F, Paal M, Mikus G, Vogeser M, Habler K, Huisinga W, Zoller M, Michelet R, Kloft C, Liebchen U. Model-informed identification of optimised dosing strategies for meropenem in critically ill patients receiving SLEDD: an observational study. Infection. 2025 Oct;53(5):1819-1831. doi: 10.1007/s15010-025-02504-0. Epub 2025 Apr 25. PMID 40279026
- [Derived] Scharf C, Weinelt F, Schroeder I, Paal M, Weigand M, Zoller M, Irlbeck M, Kloft C, Briegel J, Liebchen U. Does the cytokine adsorber CytoSorb(R) reduce vancomycin exposure in critically ill patients with sepsis or septic shock? a prospective observational study. Ann Intensive Care. 2022 May 23;12(1):44. doi: 10.1186/s13613-022-01017-5. PMID 35599248
- [Derived] Scharf C, Liebchen U, Paal M, Taubert M, Vogeser M, Irlbeck M, Zoller M, Schroeder I. The higher the better? Defining the optimal beta-lactam target for critically ill patients to reach infection resolution and improve outcome. J Intensive Care. 2020 Nov 23;8(1):86. doi: 10.1186/s40560-020-00504-w. PMID 33292582